CLINICAL TRIAL: NCT07010107
Title: Efficacy and Safety of Anaprazole in the Treatment of Reflux Esophagitis: A Multicenter, Randomized, Double-Blind, Double-Dummy, Parallel-Group, Positive-Controlled Phase III Clinical Trial.
Brief Title: A Clinical Trial of Anaprazole for Treating Reflux Esophagitis.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Xuanzhu Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3571-RE-3001
Record Dates: First submitted 2025-05-30; First posted 2025-06-08 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Reflux Esophagitis (RE)
Keywords: Anaprazole; Rabeprazole; Reflux Esophagitis
MeSH Terms: conditions — Esophagitis, Peptic | interventions — Rabeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anaprazole (Experimental): Anaprazole 3 tablets (20 mg/tablet) + Rabeprazole placebo 1 tablet (0.16 g/tablet), administered orally 30-60 minutes before breakfast once daily for up to 8 weeks. After 4 weeks of continuous treatment, if endoscopic evaluation confirms the cure of reflux esophagitis, treatment may be discontinued.
  Interventions: Drug: Anaprazole + Rabeprazole placebo
- Rabeprazole (Active Comparator): Rabeprazole 1 tablet (20 mg/tablet) + Anaprazole placebo 3 tablets (0.2 g/tablet), orally administered 30-60 minutes before breakfast once daily for up to 8 weeks. After 4 weeks of continuous treatment, if endoscopic evaluation confirms the cure of reflux esophagitis, treatment may be discontinued.
  Interventions: Drug: Rabeprazole + Anaprazole placebo

INTERVENTIONS:
Drug: Anaprazole + Rabeprazole placebo — Anaprazole 3 tablets (20 mg/tablet) + Rabeprazole placebo 1 tablet (0.16 g/tablet), administered orally 30-60 minutes before breakfast once daily for up to 8 weeks. After 4 weeks of continuous treatment, if endoscopic evaluation confirms the cure of reflux esophagitis, treatment may be discontinued.
  Arms: Anaprazole
Drug: Rabeprazole + Anaprazole placebo — Rabeprazole 1 tablet (20 mg/tablet) + Anaprazole placebo 3 tablets (0.2 g/tablet), orally administered 30-60 minutes before breakfast once daily for up to 8 weeks. After 4 weeks of continuous treatment, if endoscopic evaluation confirms the cure of reflux esophagitis, treatment may be discontinued.
  Arms: Rabeprazole

SUMMARY:
This Phase III clinical trial is designed to assess the efficacy and safety of Anaprazole 60 mg once daily (QD) administered over a period of up to 8 weeks, compared with Rabeprazole 20 mg QD, in patients with reflux esophagitis.

ELIGIBILITY:
Inclusion Criteria:

1. The patients provided voluntary signed informed consent forms.
2. Aged ≥18 years and ≤75 years old.
3. Endoscopically diagnosed as reflux esophagitis (LA grade B-D) within 14 days before randomization.

Exclusion Criteria:

1. Researchers believe that patients with uncontrolled primary diseases are not suitable for clinical trials, particularly those with a history of severe conditions affecting the cardiovascular, nervous, respiratory, hepatic, renal, or other systems.
2. Patients with concomitant diseases that may affect the esophagus or esophageal motility and, could potentially influence the efficacy evaluation.
3. Patients with a history of prior surgical procedures that could potentially impact esophageal function, or surgeries.
4. Patients confirmed to have active peptic ulcers or active upper/lower gastrointestinal bleeding within the last 30 days via esophagogastroduodenoscopy (EGD).
5. Patients with a history of Zollinger-Ellison syndrome, achalasia of the cardia, secondary esophageal motility disorders, irritable bowel syndrome, inflammatory bowel disease, or other gastrointestinal functional disorders.
6. Patients with a history of malignant tumor or having received treatment for malignant tumor within 5 years prior to randomization.
7. Patients with a history of mental illness or a history of drug or alcohol abuse within 12 months prior to screening.
8. Patients who tested positive for HIV, HBsAg, and/or HCV antibodies during screening.
9. Patients with malignant tumors or a predisposition to malignancy in the stomach or esophagus.
10. Patients with abnormal liver function: AST and/or ALT levels ≥2.0×ULN, and/or total bilirubin (TBIL) levels ≥1.5×ULN.
11. Patients with abnormal renal function: Serum creatinine levels ≥1.5×ULN, blood urea or blood urea nitrogen levels ≥1.5×ULN.
12. Patients with clinically significant ECG abnormalities, including QTc interval prolongation (QTcF ≥450 ms for men and QTcF ≥470 ms for women).
13. Patients with poorly controlled diabetes or hypertension.
14. Patients who were unable to undergo esophagogastroduodenoscopy (EGD).
15. Patients with a known allergy to the components or ingredients of Anaprazole or Rabeprazole.
16. Patients who had used proton pump inhibitors at therapeutic doses within 14 days prior to randomization.
17. Patients who had used therapeutic doses of other drugs for treating acid reflux within 7 days prior to randomization.
18. Patients required to continue receiving non-steroidal anti-inflammatory drugs (NSAIDs), systemic glucocorticoids, or clopidogrel during the trial period.
19. Patients whose assessment may be affected by alcohol, drug, or medication withdrawal during the study.
20. Pregnant or lactating women, as well as patients planning to conceive within 30 days before randomization and up to 6 months following the trial completion.
21. Patients who had participated in other drug clinical trials within 3 months prior to randomization.
22. Patients with other conditions deemed by the researchers as unsuitable for participation in this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
The endoscopic healing rate of reflux esophagitis | Up to 8 weeks
  The endoscopic healing rate of reflux esophagitis is defined as the proportion of patients with reflux esophagitis who achieve complete mucosal healing. Complete healing is determined by the absence of mucosal breaks upon endoscopic evaluation post-treatment, and the lesion is classified as normal according to the LA classification.

SECONDARY OUTCOMES:
The endoscopic healing rate of reflux esophagitis | Up to 4 weeks
  The endoscopic healing rate of reflux esophagitis is defined as the proportion of patients with reflux esophagitis who achieve complete mucosal healing. Complete healing is determined by the absence of mucosal breaks upon endoscopic evaluation post-treatment, and the lesion is classified as normal according to the LA classification.
Changes in the severity and frequency of heartburn compared to the baseline | Up to 8 weeks
  The analysis was performed using a symptom assessment questionnaire. On Day 1 of treatment, participants reported their symptoms experienced during the 7 days prior to randomization. On Days 29 and 57 of treatment, and visits for early trial withdrawal, symptom data were recorded based on the completion status of the 7-day diary cards filled out by participants immediately preceding each visit. The severity of heartburn was evaluated using a 4-point scale, while the frequency of occurrence of heartburn was assessed using a 5-point scale.
Changes in the severity and frequency of reflux compared to the baseline | Up to 8 weeks
  The analysis was performed using a symptom assessment questionnaire. On Day 1 of treatment, participants reported their symptoms experienced during the 7 days prior to randomization. On Days 29 and 57 of treatment, and visits for early trial withdrawal, symptom data were recorded based on the completion status of the 7-day diary cards filled out by participants immediately preceding each visit. The severity of reflux was evaluated using a 4-point scale, while the frequency of occurrence of reflux was assessed using a 5-point scale.
The rate of improvement in the severity and frequency of heartburn | Up to 8 weeks
  Standard for evaluating improvement in severity of individual symptoms: Calculate the average severity score for the 7 days prior to the 4-week and 8-week visits separately. The average score = total of individual scores recorded within 7 days / number of recording days.
  * Complete remission: The average score drops to 0 points
  * Improvement: The average score decreases by at least 1 point
  * No effect: The average score remains unchanged or increases. Standard for scoring the frequency of individual symptoms: 0 points: 0 days; 1 point: 1 day; 2 points: 2-3 days; 3 points: 4-5 days; 4 points: 6-7 days; The improvement rate of individual symptom severity/frequency = (Number of improved cases / Total number of cases) × 100%.
The rate of improvement in the severity and frequency of reflux | Up to 8 weeks
  Standard for evaluating improvement in severity of individual symptoms: Calculate the average severity score for the 7 days prior to the 4-week and 8-week visits separately. The average score = total of individual scores recorded within 7 days / number of recording days.
  * Complete remission: The average score drops to 0 points
  * Improvement: The average score decreases by at least 1 point
  * No effect: The average score remains unchanged or increases. Standard for scoring the frequency of individual symptoms: 0 points: 0 days; 1 point: 1 day; 2 points: 2-3 days; 3 points: 4-5 days; 4 points: 6-7 days; The improvement rate of individual symptom severity/frequency = (Number of improved cases / Total number of cases) × 100%.
Change from baseline in the Gastroesophageal Reflux Disease Health-Related Quality of Life Questionnaire (GERD-HRQL) score | Up to 8 weeks
  GERD related quality of life (QoL) is assessed with the "gastroesophageal reflux disease - health related quality of life" (GERD-HRQL) questionnaire. QoL is measured at baseline, Days 29 and 57 of treatment, and visits for early trial withdrawal. The scale contains 10 questions and a symptom control satisfaction survey, which focuses on heartburn, acid reflux, swallowing function, and drug efficacy. Each question is scored according to a 6-point scoring criterion (0 indicates no symptoms, 5 indicates intolerable symptoms, and affects daily activities), and the total score is the sum of the scores of each item (0-50 points in total), with higher scores indicating worse quality of life. Satisfaction is divided into three levels: dissatisfaction, moderate, and satisfaction. Change in GERD-HRQL score = total GERD-HRQL score after treatment - total GERD-HRQL score before treatment.
Adverse events | Up to 8 weeks
  The treatment-emergent adverse events are evaluated by CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Changhai Hospital, Shanghai, Shanghai Municipality, China